CLINICAL TRIAL: NCT05019950
Title: A Randomized, Placebo-Controlled, Double-Blind, Single-Center Study to Evaluate Safety Tolerability and Pharmacokinetics of Oral NIM-1324 in Healthy Adult Male and Female Volunteers
Brief Title: Safety Tolerability and Pharmacokinetics of Oral NIM-1324 in Healthy Adult Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NImmune Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LABP-104-1a
Record Dates: First submitted 2021-08-16; First posted 2021-08-25 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Normal Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NIM-1324 (Experimental): Once daily oral tablet
  Interventions: Drug: NIM-1324
- Placebo (Placebo Comparator): Once daily oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NIM-1324 — Once daily oral tablet
  Arms: NIM-1324
Drug: Placebo — Once daily oral tablet
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, ascending dose, multi-cohort study. The primary objective of this study is to assess the safety and tolerability of single and 7-day repeat oral doses NIM-1324 in healthy adult volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects;
2. Adult males and females, 18 to 64 years of age (inclusive) at screening;
3. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Key Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or surgery within the past 3 months determined by the PI to be clinically relevant;
2. Current infection that requires antibiotic, antifungal, antiparasitic or antiviral medications;
3. COVID-19: Testing positive for COVID-19, a current symptomatic infection within 20 days, or an asymptomatic infection within 6 weeks.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 1 to 14 days

SECONDARY OUTCOMES:
PK | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No